CLINICAL TRIAL: NCT06556589
Title: Collaborative Care for Treatment of Depression and Anxiety
Status: Recruiting | Type: Observational
Sponsor: Kaiser Permanente (Other)
Collaborators: Garfield Memorial Fund (Other)
Responsible Party: Sponsor
Other Study IDs: 2066851; RNG212361 (Other: Kaiser Permanente Colorado)
Record Dates: First submitted 2024-07-12; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Depression; Anxiety
Keywords: Collaborative Care; Depression; Anxiety; Evaluation
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Collaborative Care offered: Implement collaborative care in at least 2 clinic locations for patients with depression and/or anxiety using population-based outreach using electronic health record tools and provider referral, and tracking outcomes in the medical record.
  Interventions: Behavioral: Collaborative Care
- No Collaborative Care offered: Provide care as usual for patients with depression and/or anxiety at all other KPCO clinics.

INTERVENTIONS:
Behavioral: Collaborative Care — Collaborative care components include patient-centered team care, population-based care, measurement-based treatment to target, evidence-based care, and accountable care.
  Groups: Collaborative Care offered

SUMMARY:
The goal of this project is to evaluate the effectiveness of a collaborative care model for primary care patients at Kaiser Permanente Colorado (KPCO) with depression and/or anxiety. Collaborative care uses evidence-based short-term treatments delivered to patients over the phone. We will explore the use of cost-efficient automated processes for patient outreach and follow-up, such as care pools of patients and using patient portal messaging, risk-based results routing to providers, and electronic health record (EHR) tools for patient tracking and outcome assessment. Using a cluster randomized design, we will compare results between clinics that are offering collaborative care to those that are not.

DETAILED DESCRIPTION:
We will answer the question: does a collaborative care model in primary care clinics improve outcomes for patients with depression and/or anxiety? Specific components of the model include:

* Patient-centered team care - virtual care management to support patient outreach, follow-up, and navigation to appropriate care settings, based on patient risk. Shared care plans with primary care and behavioral health providers, with a focus on patient preferences (e.g., short-term therapy, medications, or both) and fostering engagement in treatment.
* Population-based care - Automated workflows for population-based outreach with the Patient Health Questionnaire 9-item (PHQ9) and Generalized Anxiety Disorder 7-item (GAD7) questionnaires after diagnosis and treatment initiation for more accurate and comprehensive assessment of patient improvement. This also includes automating risk-based routing of PHQ9 results to the collaborative care team to triage patients into the most appropriate care settings and developing similar automated risk-based routing procedures for GAD7 results.
* Measurement-based treatment to target - provide short-term psychotherapy and/or pharmacotherapy with a focus on measuring treatment response with the PHQ9 and/or GAD7 to guide treatment adjustments.
* Evidence-based care - provide short-term Problem-Solving Treatment-Primary Care (PST-PC), Behavioral Activation (BA), and/or medications shown to be effective for patients in primary care settings. These evidence-based interventions will include patient engagement strategies and be applicable to diverse patient populations.
* Accountable care - The collaborative care provider team will be accountable for quality of care and clinical outcomes for the patients they serve, not just the volume of care provided.

A cluster randomized design will be used to compare depression and anxiety outcomes for at least two randomly selected KPCO primary care clinics that implement collaborative care to those clinics that provide care as usual. This design will allow us to study the effectiveness of the collaborative care model and its potential for dissemination across Kaiser Permanente regions.

ELIGIBILITY:
Inclusion Criteria:

* 18+
* Current membership and active on patient portal
* Depression Diagnosis in the prior year
* Overdue for PHQ9 Screening based on the following criteria:

  * High Risk: Last PHQ9 screener was completed greater than 4 months ago AND total Score is greater than or equal 10 or item 9 is greater than 0.
  * Low Risk: Last PHQ9 screener was completed greater than 12 months ago AND Last PHQ9 Total Score is less than 10 and item 9 is equal to 0.
* Anxiety diagnoses in the prior year
* Has a baseline GAD7 in the same prior year; score = 10+ (*Note: Provider referrals could be GAD7 score of 7 or higher)
* No Behavioral Health (BH) engagement in the prior year
* Patient is not in a Skilled Nursing Facility or Hospice
* Patient has no record of psychiatric hospitalization in the last year
* Patient does not need an interpreter (i.e., English speaking)
* Primary care location is one of the intervention clinics

Exclusion Criteria:

• Exclude individuals with any of the following diagnoses:

* Psychosis
* Dementia
* Bipolar
* Personality Disorders
* Post Traumatic Stress Disorder (PTSD)
* Obsessive Compulsive Disorder (OCD)
* Panic Disorder
* Cognitive Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with depression and/or anxiety.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9-item (PHQ-9) score | Baseline and up to 24 weeks
  Change in Patient Health Questionnaire 9-item (PHQ-9) scores before and after Collaborative Care intervention. The score ranges from 0 to 27, with lower numbers indicating improvement in depression symptoms.
Generalized Anxiety Disorder 7-item (GAD-7) | Baseline and up to 24 weeks
  Generalized Anxiety Disorder 7-item (GAD-7) questionnaire scores before and after Collaborative Care intervention. The score ranges from 0 to 21, with lower numbers indicating improvement in anxiety symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No